CLINICAL TRIAL: NCT06043284
Title: A Retrospective Study to Evaluate Verbal Scores of Children Diagnosed With Autism Spectrum Disorder Who Received Hyperbaric Treatment and Those Who Did Not Receive Hyperbaric Treatment
Brief Title: Study to Compare Verbal Scores of Children Diagnosed With ASD Who Received Hyperbaric Treatment To Those Who Did Not
Status: Completed | Type: Observational
Sponsor: Oxford Recovery Center (Other)
Collaborators: The Oxford Center (Unknown)
Responsible Party: Principal Investigator, Tami Peterson PhD, Principal Investigator, Oxford Recovery Center
Other Study IDs: OxRS-01-2021
Record Dates: First submitted 2023-06-05; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Hyperbaric Oxygen Therapy
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- HBO Treatment Group: Children diagnosed with autism spectrum disorder received applied behavior therapy and hyperbaric oxygen therapy
  Interventions: Device: Hyperbaric Oxygen Therapy
- Control Group: Children diagnosed with autism spectrum disorder received applied behavioral therapy

INTERVENTIONS:
Device: Hyperbaric Oxygen Therapy — Subjects received 100% medical grade oxygen for 60 minutes at 2.0 ATA for 40 sessions in a hard-sided monoplace hyperbaric chamber
  Groups: HBO Treatment Group

SUMMARY:
A child's ability to effectively communicate with peers, parents, and caregivers impacts their level of independence and quality of personal relationships. This retrospective study will compare the speech development of participants aged 2 - 17 years that received 40 sessions of HBOT at 2.0 ATA to those who had not. Both groups will have a verbal assessment every six months. There were 32 subjects in the HBO group and 33 subjects in the non-HBO group. The statistical analysis will focus on whether Hyperbaric Oxygen Therapy made a significant difference in Verbal Behavior Milestones Assessment and Placement Program (VB-MAPP) or Assessment of Basic Language and Learning Skills (ABLLS) results.

DETAILED DESCRIPTION:
Methods: This was a study designed to retrospectively determine any association between hyperbaric oxygen therapy (HBOT) and change in verbal scores in children with autism spectrum disorder (ASD). All children aged 2 to 17 years, diagnosed with ASD who completed a verbal test every six months (either Verbal Behavior Milestones Assessment and Placement Program or the Assessment of Basic Language and Learning Skills), received applied behavioral analysis at Oxford Recovery Center (ORC) were screened for inclusion, some of whom had elected to receive HBOT (at least 40 sessions for 60 minutes at 2.0 ATA).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with autism spectrum disorder by a qualified practitioner
* Obtained medical clearance for hyperbaric oxygen therapy
* Received applied behavioral analysis at Oxford Recovery Center
* Received two of the same age appropriate verbal test 6 months apart

Exclusion Criteria:

* History of seizure disorder
* Diagnosis of genetic or mitochondrial mutation

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The medical records were reviewed for children aged 2 - 17 years who were diagnosed by a qualified practitioner with autism spectrum disorder (ASD) and treated at the Oxford Recovery Center between Jan 2018 and July 2021. Each child who underwent a minimum of 40 hyperbaric oxygen treatments at 2.0 ATA in a hard sided monoplace chamber, had two age-appropriate verbal tests 6 months apart, and received applied behavioral analysis during the study period were included in the treatment group. Children who did not undergo hyperbaric oxygen therapy, received two age-appropriate verbal tests 6 months apart, and received applied behavioral analysis were included in the control group. Any child diagnosed with seizure disorder, genetic or mitochondrial mutation were excluded from the study cohort.
Sampling Method: Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-02-20 (Actual)

PRIMARY OUTCOMES:
The verbal scores will be measured for children with autism who underwent hyperbaric oxygen therapy and compared to those who did not by an age appropriate assessment. | Change from baseline of verbal scores at 6 months
  Verbal testing: Verbal Behavior Milestones Assessment and Placement Program (VBMAPP)
The verbal scores will be measured for children with ASD who underwent hyperbaric oxygen therapy and compared to the those who did not using an age appropriate assessment. | Change from baseline of verbal scores at 6 months
  Verbal testing: Assessment of Basic Language and Learning Skills (ABLLS).

SECONDARY OUTCOMES:
Number of participants with hyperbaric oxygen treatment related adverse events. | up to 30 weeks
  Adverse events were collected during every HBO session only for the treatment group subjects. All verbatim AE terms were coded using the Medical Dictionary for Regulatory Activities (MedDRA) and summarized by system organ class (SOC) and, preferred term (PT) and study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sherwin, MD, Study Director — Wayne State University
Locations (2):
- United States (2):
  - Oxford Recovery Center, Brighton, Michigan
  - Oxford Recovery Center, Troy, Michigan

IPD SHARING:
Plan to Share IPD: Yes